CLINICAL TRIAL: NCT05164705
Title: Improving Human Cerebrovascular Function Using Acute Intermittent Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Molly Bright, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00215559
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Healthy Brain Perfusion
Keywords: Acute Intermittent Hypoxia; MRI; Perfusion; Cerebral Blood Flow; Cerebrovascular Reactivity

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled crossover trial
Who Masked: Participant
Masking Description: Participants will not know whether they are receiving active or sham hypoxia during individual AIH sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Hypoxia (Active Comparator): Participant will visit our center 2-4 times per week for three weeks to receive Acute Intermittent Hypoxia.
  Interventions: Other: Acute Intermittent Hypoxia
- Sham Intermittent Hypoxia (Sham Comparator): Participants will visit our center 2-4 times per week for three weeks to receive Sham Intermittent Hypoxia.
  Interventions: Other: Sham Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — Participants will wear a non-rebreathing face mask and alternate between breathing 9% O2 gas mixture for up to 1 minute, or until the target SpO2 of 85 percent is reached, and normal room air (21 percent O2) until 2 minutes are complete. This cycle will be repeated 15 times, resulting in a 30-minute protocol.
  Arms: Intermittent Hypoxia
Other: Sham Acute Intermittent Hypoxia — Participants will wear a non-rebreathing face mask and breathe normal air (21 percent O2) for 30-minutes.
  Arms: Sham Intermittent Hypoxia

SUMMARY:
This study uses magnetic resonance imaging to determine whether 3 weeks of repeated exposure to Acute Intermittent Hypoxia can improve brain blood flow or blood flow regulation in healthy adults.

DETAILED DESCRIPTION:
This study aims to identify an intervention to improve the function of blood vessels in the human brain, in order to mitigate damage to overall brain function and improve health outcomes across the lifespan. Hypoxia is a potent driver of angiogenesis and vascular plasticity, and acute intermittent hypoxia (AIH) protocols, in which an individual alternates between breathing mildly hypoxic air and normal air, are being rigorously examined for their potential in improving human physiology. This study tests whether AIH evokes beneficial vascular plasticity in the human brain, using a randomized crossover design to determine the impact of different daily AIH or sham interventions on MRI measures of cerebrovascular physiology.

Healthy, able-bodied participants between 21 and 50 years old will be invited to participate in this study. The daily AIH intervention consists of repeated visits to the PI laboratory over a three-week period to have an AIH or sham protocol administered via a hypoxia generator and face mask (Hyp-123, Hypoxico). Blood pressure readings will be taken before and after all intervention visits, and SpO2 levels continuously recorded for safety monitoring.

The effectiveness of the different interventions at improving cerebrovascular function will be assessed using MRI. In the week prior to each intervention period the participant will undergo MRI scanning. In addition to structural and diffusion weighted scans, multiple perfusion metrics will be extracted. Whole-brain cerebral blood flow will be measured using phase-contrast MRI, and quantitative CBF maps of regional perfusion will be measured using arterial spin labeling MRI. These perfusion metrics will be acquired three times: during normoxic (baseline), hypoxic, and hypercapnic conditions. Changes in perfusion values during gas challenges will measure whole-brain and regional cerebrovascular reactivity. The MRI protocol will be repeated one day after the last intervention visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between ages of 21 and 50 years
* No known neurological, respiratory or vascular conditions
* Safe to be scanned using MRI
* Able to communicate in English

Exclusion Criteria:

* MRI contraindications as indicated on MRI safety screening form
* Subjects with pacemakers, cochlear (in the ear) implants, or aneurysm clips or subjects who have worked with metal
* Pregnant women
* Individuals with known neurological or vascular conditions
* Individuals with sleep apnea, emphysema, or other respiratory conditions
* Individuals with severe claustrophobia
* Subjects unwilling or unable to give written informed consent in English
* Prisoners
* Frequent smoker
* Allergy to Tegaderm
* Blood pressure greater than 140/90 or less than 90/55.
* Individuals who report headaches, feeling dizzy or light-headed, or have heart palpitations on the day of the study.
* Individuals prescribed Aripiprazole and/or Lamotrigine*

Note, mild (well-controlled) asthma is not immediate grounds for exclusion.

*Other prescription medications may be grounds for exclusion; prescription medication information will be acquired during initial screening and at subsequent follow-up visits

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Resting cerebral blood flow | 4 weeks
  Phase-contrast MRI and Arterial Spin Labeling MRI will be used to quantify whole-brain and cortical gray matter perfusion (ml/100g/min) before and after the 3-week intervention.

SECONDARY OUTCOMES:
Cerebrovascular reactivity | 4 weeks
  Phase-contrast MRI and Arterial Spin Labeling MRI will be used to quantify the change in perfusion caused by a vasodilatory gas challenge (inhaled hypoxia or hypercapnia), before and after the 3-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Molly G Bright, DPhil, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
MR imaging data and the associated physiologic data collected during MRI scanning will be shared in an anonymized format, along with the extracted quantitative perfusion maps and cerebrovascular reactivity maps. These data will be made available to public through the Open Science Framework (osf.io) or similar public repository. Code will be made available through the PI's laboratory Github account. A link to these resources will be included with publications resulting from this study to facilitate access.
Supporting Information: Analytic Code
Time Frame: At time of publication (or within one year of project completion, whichever occurs first).
Access Criteria: Data will be anonymized and made publicly available, and at that time no approval is needed and therefore there are no access criteria.

REFERENCES:
- [Derived] Johnson HR, Wang MC, Stickland RC, Chen Y, Parrish TB, Sorond FA, Bright MG. Variable cerebral blood flow responsiveness to acute hypoxic hypoxia. Front Physiol. 2025 Mar 12;16:1562582. doi: 10.3389/fphys.2025.1562582. eCollection 2025. PMID 40144550

DOCUMENTS (1):
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT05164705/ICF_001.pdf